CLINICAL TRIAL: NCT04253353
Title: A PHASE 1, OPEN LABEL, TWO-PERIOD, TWO-TREATMENT, FIXED-SEQUENCE STUDY TO ESTIMATE THE EFFECT OF A MULTIPLE ORAL DOSE OF TAFAMIDIS ON ROSUVASTATIN PHARMACOKINETICS IN HEALTHY PARTICIPANTS
Brief Title: A Drug-Drug Interaction Study To Estimate The Effect Of Tafamidis On Rosuvastatin Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B3461075
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tafamidis; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rosuvastatin and tafamidis fixed sequence (Experimental): * Period 1: rosuvastatin 10 mg (single oral administration)
  * Washout
  * Period 2: tafamidis 61 mg capsule(multiple doses, twice a day) + rosuvastatin 10 mg (single oral administration)
  Interventions: Drug: tafamidis; Drug: rosuvastatin

INTERVENTIONS:
Drug: tafamidis — 61 mg capsule
  Other Names: Vyndaqel
Drug: rosuvastatin — 10 mg tablet
  Other Names: Crestor

SUMMARY:
Each subject will be given a single oral dose of rosuvastatin on Day 1 in Period 1. In Period 2, after a washout period of at least 5 days, each subject will receive oral doses of tafamidis twice daily (BID) on days 1 and 2, followed by tafamidis once daily (QD) on days 3 to 9 with an oral dose of rosuvastatin on Day 7. Rosuvastatin exposures will be compared between Periods 1 and 2 to estimate the effect of tafamidis on rosuvastatin PK in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 60 years of age, inclusive, at the time of signing the informed consent document (ICD)
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiovascular tests
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* History of hypersensitivity to rosuvastatin., asymptomatic, seasonal allergies at the time of dosing).
* Use of CYP2C19 inhibitors (eg, fluconazole, fluoxetine, fluvoxamine, ticlopidine omeprazole, voriconazole, cimetidine, esomeprazole, and felbamate) or inducers (eg, rifampin, ritonavir, efavirenz, enzalutamide, phenytoin, and St. John's Wort) within 28 days or 5 half-lives (whichever is longer) prior to dosing.
* Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or other inducers (eg, phenytoin, carbamazepine) within 28 days or 5 half-lives (whichever is longer) prior to dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time 0 extrapolated to infinity (AUCinf) for rosuvastatin | Hours 0, at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose in Periods 1 and 2.
  AUClast + (Clast/kel)
Apparent renal clearance (CLr) for rosuvastatin | Hours 0, at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose in Periods 1 and 2 for AUClast. For Ae, hours 0-24, 24-48, 48-72 hours post-dose in Periods 1 and 2.
  Ae/AUClast for extravascular dosing

SECONDARY OUTCOMES:
Number of subjects with a clinically significant change in vital sign measurements from baseline | Baseline through Day 10 of period 2
Number of subjects with a clinically significant change in laboratory tests from baseline | Baseline through Day 10 of period 2
Number of subjects with treatment emergent adverse events | Baseline through Day 28 follow up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461075